CLINICAL TRIAL: NCT01344044
Title: A Randomised Controlled Trial of a Brain-Computer Interface Based Intervention for the Treatment of ADHD
Brief Title: Brain-Computer Interface (BCI) Based Intervention for Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Healthcare Group, Singapore (Other Government)
Collaborators: Duke-NUS Graduate Medical School (Other); Agency for Science, Technology and Research (Other); Singapore Clinical Research Institute (Other)
Responsible Party: Principal Investigator, Lim Choon Guan, Dr, National Healthcare Group, Singapore
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DSRB Domain A/09/395
Record Dates: First submitted 2011-04-27; First posted 2011-04-28 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Brain-Computer Interface
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Brain-Computer Interfaces

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BCI treatment (Active Comparator): BCI treatment will commence during the week of the Baseline.
  Interventions: Device: BCI
- Wait-list control (Other): BCI treatment will commence 8 weeks after Baseline
  Interventions: Device: BCI
- BCI pilot arm (Experimental): This is a experimental arm to test out the safety and effectiveness of BCI in improving ADHD symptoms. This pilot arm is necessary as the BCI device, incorporating dry electrode sensors and intervention game, is newly developed and have not been tested out in children with ADHD. This preliminary study will also allow us to test out the treatment protocol (24 sessions of BCI training over 8 weeks) to see if it is efficacious.
  Interventions: Device: BCI

INTERVENTIONS:
Device: BCI — 24 half-hour sessions over 8 weeks, i.e. 3 sessions per week, followed by 3 once-monthly boosters.
  Other Names: Brain-Computer Interface

SUMMARY:
This study aims to examine the efficacy of a brain-computer interface system for the treatment of inattentive symptoms of Attention Deficit Hyperactivity Disorder (ADHD). The investigators hypothesis is that children with ADHD receiving treatment with the BCI-based training will improve to a greater extent than the control group.

Additionally, the investigators are also conducting an fMRI study involving interested participants, to elucidate the neural mechanisms underlying any behavioural improvement. This is necessary to help the investigators gain a better picture of brain correlates related to ADHD and understand how the intervention can affect the brain.

DETAILED DESCRIPTION:
This BCI study will involve 2 phases. The first phase is a preliminary study to test the safety and effectiveness of the novel BCI device which involves newly developed dry electrode sensors and intervention game. Twenty children, aged 6-12 and diagnosed with Inattentive or Combined subtype of ADHD will be recruited for the study. This open-label, experimental arm will go through 8 weeks of BCI intervention.

The second phase will be a randomized controlled trial involving 160 children. They will be randomized into the treatment or control arm. The treatment arm will receive 8 weeks of BCI intervention, similar to the experimental arm. The other group will serve as wait-list controls.

The fMRI trial aims to examine the underlying neural processes explaining any therapeutic effects that may be seen.

The study will enroll 70 children with ADHD, aged 6-12, who are participating in the main randomized controlled trial: 40 from the BrainpalTM intervention group and 30 from the control group; participants will undergo fMRI scan at Week 0 and 8 or Week 8 and 16. The study will recruit another 30 children aged 6-12 from the community as the healthy control group, who will undergo the same imaging procedure once. The scans will involve both functional and structural imaging.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-TR criteria for ADHD, either the combined or inattentive subtype, based on the Diagnostic Interview Schedule for Children (CDISC; Schaffer et al., 2000)

Exclusion Criteria:

* Present or history of medical treatment with stimulant medication and Atomoxetine
* Co-morbid severe psychiatric condition or known sensori-neural deficit e.g. complete blindness or deafness (such that they cannot play computer games)
* History of epileptic seizures
* Known Developmental Delay (i.e. IQ 70 and below)
* Predominantly Hyperactive/impulsive subtype of ADHD (i.e. no predominant inattentive symptoms)
* Present/history polyunsaturated fatty acids supplement intake (e.g. Omega-3 oil, flax seed oil, cod liver oil) in the past 3 months
* Present/history of traditional Chinese medicine (TCM) prescribed for treatment of attention problems in the past 1 month

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2011-01; Primary Completion 2016-05-13 (Actual); Study Completion 2016-05-13 (Actual)

PRIMARY OUTCOMES:
Attention Deficit Hyperactivity Disorder Rating Scale (ADHD Rating Scale) 4th Edition | Week 0, 8, 20, 24

CONTACTS AND LOCATIONS:
Overall Officials: Choon Guan Lim, Principal Investigator — Institute of Mental Health, Singapore
Locations (1):
- Child Guidance Clinic, Institute of Mental Health, Singapore, Singapore

REFERENCES:
- [Derived] Lim CG, Soh CP, Lim SSY, Fung DSS, Guan C, Lee TS. Home-based brain-computer interface attention training program for attention deficit hyperactivity disorder: a feasibility trial. Child Adolesc Psychiatry Ment Health. 2023 Jan 25;17(1):15. doi: 10.1186/s13034-022-00539-x. PMID 36698168
- [Derived] Lim CG, Lee TS, Guan C, Fung DS, Zhao Y, Teng SS, Zhang H, Krishnan KR. A brain-computer interface based attention training program for treating attention deficit hyperactivity disorder. PLoS One. 2012;7(10):e46692. doi: 10.1371/journal.pone.0046692. Epub 2012 Oct 24. PMID 23115630